CLINICAL TRIAL: NCT05855850
Title: DIfferential Feasibility and Tolerability of Deep repetitiVe transcranIal MagNEtic Stimulation for Depression in Older Adults (DIVINE Trial): A Pilot Study
Brief Title: Deep rTMS for Depression in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Peter Boris Centre for Addictions Research (PBCAR) (Unknown)
Responsible Party: Principal Investigator, Dante Duarte, Principal Investigator, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15344
Record Dates: First submitted 2023-02-06; First posted 2023-05-12 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD; depressive disorder; depression; late-life depression; mood disorders; deep transcranial magnetic stimulation; deep TMS; dTMS; H coil; H-coil; older adults; H4-coil; H7-coil
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder; Depression; Mood Disorders

STUDY DESIGN:
Intervention Model Description: This investigation is a one-way two-group between-subjects open-label design
Masking Description: This is an open label trial. Only study staff processing and analyzing the data will be fully blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active H4-coil dTMS treatment (Experimental)
  Interventions: Device: Brainsway H4-Coil Deep TMS System
- Active H7-coil dTMS treatment (Experimental)
  Interventions: Device: Brainsway H7-Coil Deep TMS System

INTERVENTIONS:
Device: Brainsway H4-Coil Deep TMS System — Participants assigned to this arm will complete a 4-week course of 5 dTMS sessions per week (using the Brainsway H4-coil), for a total of 20 stimulation sessions. We will follow the standard Health Canada and FDA-approved protocol for depression: 18 Hz and 55 trains, for a total of 1980 pulses.
  Arms: Active H4-coil dTMS treatment
Device: Brainsway H7-Coil Deep TMS System — Participants assigned to this arm will complete a 4-week course of 5 dTMS sessions per week (using the Brainsway H7-coil), for a total of 20 stimulation sessions. We will follow the standard Health Canada and FDA-approved protocol for depression: 18 Hz and 55 trains, for a total of 1980 pulses.
  Arms: Active H7-coil dTMS treatment

SUMMARY:
This study aims to: (1) assess the feasibility and tolerability of two active dTMS coils - H4 and H7 - in older adults with depression; and (2) clinical response measured by change from baseline on the Hamilton Depression Rating Scale- 24 item; changes in cognitive function through neuropsychological assessment; and changes in regional electrophysiological activity and functional connectivity indexed by EEG. Through a parallel design, participants will complete a four-week course of five dTMS sessions per week, for a total of 20 stimulation sessions. Participants will be randomly assigned to either coil (H4 or H7) and will complete questionnaires examining side effects, mental health symptoms, and cognition. Participant EEG data will be measured and collected at baseline and at the end of each week. Collectively, the study will address the absolute and differential feasibility and tolerability of the two active coils to provide preliminary data for a future randomized controlled trial comparing one or both of these novel interventions to the established H1-coil and a sham stimulation (placebo) control.

DETAILED DESCRIPTION:
Transcranial magnetic stimulation (TMS) is a non-invasive therapeutic technique used to stimulate regions of the brain using magnetic pulses. Repeated TMS delivers sequences of pulses for multiple days in a row and is an approved treatment for several psychiatric conditions. Deep TMS (dTMS) is a new technique that uses modified magnetic Hesed coils (H-coils) to stimulate deeper regions of the brain and has been FDA- and Health Canada-approved for major depressive disorder (MDD), obsessive-compulsive disorder, smoking cessation, and anxious-depression in adults. For older adults (60+), traditional rTMS has also shown efficacy for MDD (60+) and one RCT has found benefit for the H1 dTMS coil, but no trials have examined the H4 and H7 coils in this population. This innovative pilot study will explore dTMS feasibility and tolerability (i.e., side effects, impacts on mental health and cognition) of these two dTMS coils (H4, targeting insula and H7, targeting anterior cingulate cortex) in older adults with depression. The pilot will provide critical preliminary data for a future trial comparing these novel interventions to the H1-coil and a sham stimulation control. There is sparse literature examining the effects of dTMS on cognition, as measured by neuropsychological testing, and brain activity, as measured by electroencephalogram (EEG), while comparing different dTMS H-coils. Therefore, a second feature of the design includes assessing both domains over the course of treatment. The results will lay the foundation for a future randomized controlled trial examining the efficacy and mechanisms of one or both of these novel forms of neurostimulation for MDD in older adults.

ELIGIBILITY:
Inclusion Criteria:

A) 60 - 85 years old

B) Able to provide informed consent to participate in the study

C) MDD diagnosis, single or recurrent episode, assessed using Evaluation of the Diagnostic Assessment Research Tool (DART) Screener for DSM-5 Mood Disorder Module

D) Total score of at least 20 on the 24-item Hamilton Depression Rating Scale (HDRS-24) at screening visit

E) Treatment resistance to antidepressant pharmacotherapy during the current episode as indexed by Antidepressant Treatment History Form - Short Form (ATHF - SF). Specifically, participants will be required to have failed at least one or to have had an inadequate trial (including intolerance) to at least two antidepressants in the current episode

F) Participants will be required to be on stable dosages of other psychotropic medications for at least 4 weeks prior to screening

Exclusion Criteria:

A) Primary diagnosis of bipolar I or II disorder; psychotic disorder; obsessive-compulsive, post-traumatic stress, anxiety, or personality disorder; participants with anxiety or personality disorders will be eligible if is not their primary diagnosis

B) Active suicidal behavior

C) Substance dependence/abuse in the past 3 months before entering the study (this will be screened via self-report and verified by urine screening test)

D) Possible dementia diagnosis based on a Mini Mental Status Exam (MMSE) score of <24 and clinical presentation of dementia

E) Unsuccessful ECT treatment on the current episode

F) Traditional contraindications to rTMS: Intracranial or metal implants in the head or nearby regions, excluding the mouth, that cannot be safely removed; History of epilepsy or seizures; Active unstable medical condition (recent laboratory and neuroimaging alterations); Pacemaker and/or implantable cardioverter-defibrillators; current use of bupropion >300 mg/day as it is associated with risk of seizures, treatment with equivalent benzodiazepine dose to lorazepam >2 mg/day

G) People with severe literacy, visual, or hearing issues that affect their ability to engage in the interviews

H) People with recurring migraines or headaches (weekly or more).

I) Individuals residing beyond the borders of the Greater Hamilton Area and its neighbouring vicinities.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — We will implement a sex equity approach by aiming at a 50/50% rate of male and female but allowing an imbalance of maximum 60/40% from either side.
Enrollment: 21 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Feasibility criteria 1: Protocol completion | 4 weeks
  Percentage of intervention sessions completed
Feasibility criteria 2: Retention rate | 4 weeks
  Percentage of participants who complete study once enrolled
Feasibility criteria 3: Screening rates and capacity | 4 weeks
  Number of participants (n) screened; n enrolled as a percentage of n screened monthly
Feasibility criteria 4: Recruitment rate and capacity | 4 weeks
  Total number of participants recruited and enrolled per month.
Feasibility criteria 5: Duration of intervention and assessment processes | 4 weeks
  Compared to estimated times, the actual mean times (in min) from start to finish for each dTMS intervention session and mean time (in hours) from start to finish for each visit.
Feasibility criteria 5: Safety of H-coil dTMS treatment | 4 weeks
  Total number of adverse events reported during the treatment sessions assessed by the Side Effects Questionnaire for dTMS (custom-developed for study). At each dTMS stimulation session, participants will complete a questionnaire to evaluate potential adverse effects of dTMS (headache, neck pain, itching and redness at the site of stimulation) according to a 4-point scale.
Tolerability of H-coil dTMS treatment | 4 weeks
  Percentage of participants withdrawn or terminated following enrollment due to adverse events

SECONDARY OUTCOMES:
Change from baseline on the Hamilton Depression Rating Scale- 24 item (HDRS-24). | 4-weeks + 2-week follow-up
  The Hamilton Depression Rating Scale (24 item) will be used as the primary measure of depression. Symptoms of depression will be assessed with the HDRS- 24 item (a 24-item depression checklist) at multiple visits: the in-person screen (V0), baseline (V1), end-of-week dTMS sessions (V5, V10, V15, V20), and the 2-week follow-up. Scores range from 0 (min) to 75 (max), with a score of ≥ 20 indicating a moderate-to-severe depression. Lower scores may indicate mild depression or remission.
Changes from baseline on the Geriatric Depression 30-item Scale (GDS-30) | 4-weeks + 2-week follow-up
  The Geriatric Depression 30-item Scale (GDS-30) will be used as a second measure of depression, a 30-item checklist, at the baseline (V1), midpoint (V10) and endpoint (V20) visits and at the 2-week follow-up. Scores of 0-4 are considered normal, 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
Change from baseline on the General Anxiety Disorder- 7 item (GAD-7) | 4-weeks + 2-week follow-up
  Symptoms of anxiety will be assessed using this 7-item questionnaire at the baseline (V1), midpoint (V10) and endpoint (V20) visits and at the 2-week follow-up. Scores of 0-4 indicate minimal anxiety; 5-9: mild anxiety; 10-14: moderate anxiety; and 15 or greater: severe anxiety.
Change from baseline on the Pittsburgh Sleeping Quality Index (PSQI) | 4-weeks + 2-week follow-up
  Sleep will be monitored and assessed using the Pittsburgh Sleeping Quality Index (PSQI) at the baseline (V1), midpoint (V10) and endpoint (V20) visits and at the 2-week follow-up. Each of component of the PSQI is issued a score ranging from 0 to 3, with 3 indicating the greatest dysfunction.
Change from baseline on the Patient Health Questionnaire (PHQ - Somatic Symptoms) | 4-weeks + 2-week follow-up
  Somatic symptoms will be evaluated using the Patient Health Questionnaire (PHQ) somatic inventory at the baseline (V1), midpoint (V10) and endpoint (V20) visits and at the 2-week follow-up. Scores range from 0 to 30: ≥ 5 = mild, ≥ 10 = moderate, and ≥ 15 = severe levels of somatization.
Changes from baseline in resting-state EEG | 4 weeks
  Using electroencephalography (EEG), we will assess alpha, theta and gamma rhythms in fronto-temporo-parietal region, including assessment of connectivity and coherence. We will additionally measure cross-frequency coupling named theta (4-8Hz)-gamma (>25Hz) phase-amplitude coupling (PAC). We will also investigate phase synchronization in upper theta frequency band between prefrontal and temporal areas. Changes in these EEG parameters will be correlated with changes in mood severity and cognitive status, with a focus on working memory improvements. EEG will be performed before dTMS sessions at baseline (V1) and at the end of each week (V5, V10, V15 and V20) by using a wireless dry electrode portable EEG system (CGX Quick 20r). Resting state connectivity, coherence, PAC, and synchronization assessed by EEG will use standardized data processing pipelines in EEG Lab.
Changes from baseline in neurocognitive functioning (Repeatable Battery of Neuropsychological Status [RBANS]) | 4 weeks
  Neurocognitive performance will be assessed with the Repeatable Battery of Neuropsychological Status. Assessments will be completed at baseline (V1) and at post-treatment (V20).

CONTACTS AND LOCATIONS:
Overall Officials: Dante Duarte, MD, MSc, PhD, Principal Investigator — Peter Boris Centre for Addictions Research at St. Joseph's Healthcare, Hamilton; James MacKillop, PhD, Study Director — Peter Boris Centre for Addictions Research at St. Joseph's Healthcare, Hamilton; Emily MacKillop, PhD, ABPP-CN, Study Chair — Peter Boris Centre for Addictions Research at St. Joseph's Healthcare, Hamilton
Locations (1):
- Peter Boris Centre for Addictions Research, St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada